CLINICAL TRIAL: NCT07026019
Title: Effects Of Tele-Based Multimodal Versus Bruegger's Relief Exercise Program In Electronic Gadget Users With Chronic Mechanical Neck Pain
Brief Title: Exercise and Chronic Mechanical Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Kiran- REC/RCR&AHS 24/0139
Record Dates: First submitted 2025-06-11; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Neck Pain Chronic
Keywords: Neck pain; Telehealth; Range of motion; Photogrammetry
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal exercise program (Active Comparator)
  Interventions: Other: Multimodal exercise program
- Bruegger's Relief Exercise (Experimental)
  Interventions: Other: Bruegger's relief exercise

INTERVENTIONS:
Other: Bruegger's relief exercise — Participant will be in a high sitting position. An elastic resistance band will be wrapped on each hand of the participant leaving the palm open and will be told to abduct and extend of thumb along with fingers, followed by wrist extension and forearm supination, the participant will be instructed to perform scapular retraction with shoulder external rotation, elbow extension, shoulder abduction, and extension and chin tuck. The treatment protocol will be for 4 weeks, having 3 sessions in a week and 4 sets of 12 repetitions in each session. Intervention was started from 10 seconds hold to 30 seconds with 2 seconds increment in every session. Rest time was 30 seconds.
  Arms: Bruegger's Relief Exercise
Other: Multimodal exercise program — Multimodal exercise program including chin tucks, bilateral pectoral stretching, scapular region strengthening exercises and Wand exercises. The training program applied 3 times a week, 50 minutes each time, for 4 weeks
  Arms: Multimodal exercise program

SUMMARY:
This Randomized Clinical Trial will be conducted at Riphah Rehabilitation and Research Center and spans 4 weeks. Non-probability Convenient sampling will be used to collect the data. A sample size of 40 subjects with age group between 18-45 years will be taken. Data will be collected from patients who use electronic gadgets and have present complaints of mechanical neck pain. Outcome measures will be taken using the Numeric pain rating scale (NPRS) for pain, Neck Disability Index (NDI) for disability, Goniometer for Range of motion, and Kinovea software for shoulder, eye, and craniovertebral angle measurement. Subjects will be selected based on inclusion and exclusion criteria and will be equally divided into two groups by random number generator table. The first assessment will be conducted physically and after that, both groups will receive treatment via MS teams under the supervision of a physiotherapist. Both the Groups will receive Hot Pack, and baseline treatment (neck isometrics, upper trapezius and scalene stretches), while Group A will receive multimodal exercises (chin tucks, bilateral pectoral stretching, scapular region strengthening exercises, and Wand exercises) and Group B will receive Bruegger's relief exercise. Outcome measures will be measured at baseline and after 4 weeks. Data analysis will be done by SPSS version 25.

DETAILED DESCRIPTION:
Neck pain is defined as "activity-limiting neck pain with or without radiation to the upper limbs lasting for at least 24 hours" is a major public health concern globally due to significant direct and indirect individual and societal costs, and the negative impact on overall health, function, well-being and quality of life. Mechanical neck pain (MNP), also known as chronic non-specific neck pain, is a common musculoskeletal chronic disease . When the duration of symptoms is greater than 12 weeks of evolution, it acquires the value of chronicity, being denominated non-specific chronic neck pain . Neck pain is a prevalent medical condition affecting a vast number of individuals worldwide. Neck pain can significantly impede daily activities and even progress into a debilitating physical disability . The annual prevalence of musculoskeletal disorders in office workers is 63% and the most common sites for musculoskeletal disorders are neck (42%) and low back (34%). Between 20% and 70% of people will experience neck pain in their lifetime .

Several epidemiological studies have reported a high prevalence of neck and shoulder pain among worldwide users of handheld devices. For example, a study of 140 handheld device users at a Canadian university showed that 68% of users had neck pain, while 46% and 52% had pain in their left and right shoulders, respectively. Also, a study of 774 smartphone users at Khon Kaen University reported that 48.4% of users had shoulder pain, and 43.1% of users had neck pain. Interestingly, regarding posture when using a smartphone, it was found that 91% of 859 subjects had a flexed neck position, in which the head is bent down to look at the smartphone screen, and the head is tilted in a forward position for a long time, which causes fatigue and contributes to the development of pain in the neck. The duration of smartphone use in a poor posture for 20 minutes can induce muscle fatigue in the cervical muscles, such as the upper trapezius and cervical erector spinae muscles.

International guidelines recommend that in the absence of sinister 'red flag' pathology (e.g. fracture, neoplasm), first-line interventions for the majority of musculoskeletal conditions should involve simple non-surgical management, where interventions are tailored to the individual's needs and clinical presentation. Despite these recommendations, the timely, affordable and equitable access to such healthcare services can be severely limited for some. This has demanded organizations to rethink how traditional healthcare services can be delivered with many services rapidly adopting telehealth service delivery methods. Telerehabilitation interventions can include any type of treatment - such as treatment based on education, exercise prescription, and self-management - that can be offered at a distance. The most common ways to deliver telerehabilitation interventions are through websites, smartphone apps, videoconferences, over the telephone, and text messages.

With the growing reliance on electronic devices in daily life, understanding the most effective exercise program for managing neck pain in gadget users is essential for healthcare practitioners and individuals seeking relief. This study aims to fill a gap in current knowledge by evaluating the comparative effectiveness of tele based multimodal and Bruegger's relief exercise program, ultimately guiding healthcare professionals in recommending the most suitable exercise regimen for electronic gadget users with chronic neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Age group between 18-45 years (10).
* Both gender
* Neck pain associated with degenerative changes and myofascial pain syndromes
* Individuals having localized pain or stiffness in the cervical spine (C3-C7) without upper limb radiculopathy
* People with a disability and therefore cannot come to the clinic
* People living in highly populated cities where the healthcare system is overcrowded
* People who use electronic gadgets i.e. computers, and smartphones for more than 4 hours

Exclusion Criteria:

* Tuberculosis, carcinoma, heart disease, and osteoporosis
* Previous surgery related to the cervical spine
* Having radical symptoms such as paresis, tingling, or numbness
* Any trauma or localized infection in the neck region
* Having inflammatory rheumatologic diseases, or structural deformity
* Ongoing radiotherapy, chemotherapy, steroid therapy, or anticoagulants
* Positive Spurling's test, traction test, upper limb tension test, and shoulder abduction test

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale | Baseline, 4th Week
  The NPRS is an 11-point numeric scale in which 0 represents "NO PAIN" and 10 represents "EXTREME PAIN" (e.g., "pain as bad as you can imagine" and "worst pain imaginable").
Neck Disability Index | Baseline, 4th Week
  The NDI is a self-reported instrument for measuring perceived neck disability that consists of 10 'themes': pain intensity, personal care, weight lifting, reading, headache, concentration, work (or domestic activities), driving, sleep and recreational activities. Each question is scored from 0 to 5. The final score is expressed as a percentage
Cervical Range of Motion | Baseline, 4th Week
  Universal Goniometer, a tool used most commonly for evaluating joint ROM in the clinical settings, comes out as a simple alternative for global use at low price. Notably, the reliability and validity of cervical goniometric measurements are considered excellent, ensuring accurate measurement of cervical range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Syed Shakil ur Rehman, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Clinic, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waongenngarm P, van der Beek AJ, Akkarakittichoke N, Janwantanakul P. Perceived musculoskeletal discomfort and its association with postural shifts during 4-h prolonged sitting in office workers. Appl Ergon. 2020 Nov;89:103225. doi: 10.1016/j.apergo.2020.103225. Epub 2020 Aug 2. PMID 32755740
- [Background] Bernal-Utrera C, Gonzalez-Gerez JJ, Anarte-Lazo E, Rodriguez-Blanco C. Manual therapy versus therapeutic exercise in non-specific chronic neck pain: a randomized controlled trial. Trials. 2020 Jul 28;21(1):682. doi: 10.1186/s13063-020-04610-w. PMID 32723399